CLINICAL TRIAL: NCT02777073
Title: Effects of Single Doses of Liraglutide and Dapagliflozin on Hyperglycemia and Ketogenesis in Type 1 Diabetes
Brief Title: Effects of Single Doses of Liraglutide and Dapagliflozin on Ketogenesis in Type 1 Diabetes
Acronym: 1974
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Paresh Dandona, Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1974
Record Dates: First submitted 2015-12-01; First posted 2016-05-19 (Estimated); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Type 1 Diabetes
Keywords: Diabetic ketoacidosis; Insulin; Type 1 Diabetes; glucose (sugar) control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis; Insulin Resistance | interventions — Liraglutide; dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- liraglutide 1.8 mg (Active Comparator): single dose of Victoza ( liraglutide) 1.8 mg
  Interventions: Drug: Victoza
- Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo
- Dapagliflozin (Active Comparator): Single dose of Dapagliflozin 10 mg oral tablet
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Victoza — Single dose of Liraglutide
  Other Names: Liraglutide
  Arms: liraglutide 1.8 mg
Drug: Placebo — Single dose of generic placebo
  Arms: Placebo
Drug: Dapagliflozin 10mg Tab — single dose of 10 mg dapagliflozin
  Other Names: Dapagliflozin
  Arms: Dapagliflozin

SUMMARY:
1. To compare levels of ketone bodies (beta-hydroxybutyrate and acetoacetate) in plasma and urine following a single dose treatment of either liraglutide 1.8mg, dapagliflozin 10mg or placebo in insulinopenic state.
2. To compare plasma levels of free fatty acid, glucagon, hs-CRP, Ll-6 and IL-1 before and after administration of liraglutide/placebo.

DETAILED DESCRIPTION:
Diabetic ketoacidosis is an important cause of mortality and morbidity in type 1 patients. The decreased ratio of insulin to glucagon in insulin deficient subjects promotes ketogenesis. In patients with type 1 diabetes, the suppressive effect of hyperglycemia and the paracrine inhibitory effect of insulin and GABA from the β cell on α cell are absent. Thus, plasma glucagon concentrations are elevated and in combination with insulin deficiency, lead to lipolysis, increased plasma FFA concentrations and an increased fatty acid supply to the liver. Thus, both fatty acid oxidation and ketogenesis are enhanced.

Our recent work has shown that liraglutide, a GLP 1 agonist, improves glycemic control and reduces glycemic excursions in patients with type 1 diabetes within a few days of the initiation of treatment.

With this background, the investigators hypothesize that suppression of glucagon with liraglutide in patients with type 1 diabetes may protect them from lipolysis, increased bio-availability of FFAs, ketogenesis and ketoacidosis.

It is essential to investigate this area further as there are no prior studies that have investigated the acute effects of liraglutide on FFAs or ketogenesis. This study will be the first randomized controlled prospective study investigating the effect of liraglutide on ketogenesis. Also, it would be important to measure the mediators of inflammation at the same time to investigate whether there is a concomitant changes of inflammatory factors in parallel with the lipolysis and ketogenesis.

After the screening visit, subjects who meet the inclusion and exclusion criteria will be randomized to receive a single dose of either liraglutide, dapagliflozin or placebo and will be monitored for a total of 8 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes on continuous subcutaneous insulin infusion (CSII, also known as insulin pump).
2. Undetectable c peptide (c-peptide < 0.1 ng/ml).
3. HbA1c of less than or equal to 8.5%.
4. Age 18-75 inclusive

Exclusion Criteria:

1. Type 1 diabetes for less than 12 months
2. Coronary event/ procedure (MI, Unstable angina, CABG, PCI) in the last four weeks
3. Hepatic disease (Transaminase > 3 times normal) or Cirrhosis
4. Renal impairment (serum eGFR <30ml/min/1.73m2)
5. HIV or Hepatitis B or C positive status
6. History of pancreatitis, i.e., history of gallstones, alcohol abuse and hypertriglyceridemia
7. Pregnancy
8. Inability to give informed consent
9. History of Gastroparesis
10. Personal or Family History of medullary thyroid carcinoma or MEN 2 syndrome
11. Alcoholism
12. Hypertriglyceridemia (>500 mg/dl).
13. Those with history of bladder cancer , diabetic ketoacidosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ECMC Ambulatory Center, 3rd Floor, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin 10: single dose of Farxiga ( dapagliflozin) 10 mg
  Farxiga: Single dose of dapagliflozin
Period: Overall Study
Arm/Group | Liraglutide 1.8 mg | Dapagliflozin 10 | Placebo
Started | 13 | 17 | 13
Completed | 13 | 17 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide 1.8 mg | Dapagliflozin 10 | Placebo | Total
Number analyzed (Participants) | 13 | 17 | 13 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 13 | 43
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 7 | 24
  Male | 6 | 7 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 17 | 13 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Ketone Bodies Formation After Single Dose of Liraglutide and Dapagliflozin
Description: To compare levels of ketone bodies beta-hydroxybutyrate in plasma following a single dose treatment of either liraglutide 1.8mg,dapagliflozin 10mg or placebo in insulinopenic state.
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: mM
Groups:
- Dapagliflozin: Single dose of dapagliflozin 10 mg
Arm/Group | Liraglutide 1.8 mg | Placebo | Dapagliflozin
Number analyzed (Participants) | 13 | 13 | 17
mM | 0.08 (0.05) | 0.25 (0.05) | 0.21 (0.05)

2. Secondary Outcome: Change in Glucagon Levels.
Description: This secondary endpoint compares change in glucagon concentrations (in pg/ml) from baseline at 8 hours following liraglutide and dapagliflozin compared to placebo
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Dapagliflozin: Single dose of dapagliflozin 10mg
Arm/Group | Liraglutide 1.8 mg | Placebo | Dapagliflozin
Number analyzed (Participants) | 13 | 13 | 17
pg/mL | -19 (14) | 1 (6) | -15 (5)

3. Secondary Outcome: Change in Free Fatty Acid (FFA) Concentrations
Description: This secondary endpoint compares the change in FFA concentrations (mM) from baseline at 8 hours following liraglutide and dapagliflozin compared to placebo
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: mM
Arm/Group | Liraglutide 1.8 mg | Placebo | Dapagliflozin
Number analyzed (Participants) | 13 | 13 | 17
mM | 0.1 (0.06) | 0.17 (0.06) | 0.11 (.06)

4. Secondary Outcome: Change in Ghrelin Concentrations
Description: This secondary endpoint compares the change in ghrelin concentrations (pg/ml) from baseline at 8 hours following liraglutide and dapagliflozin compared to placebo
Time Frame: 8 Hours
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Liraglutide 1.8 mg | Placebo | Dapagliflozin
Number analyzed (Participants) | 13 | 13 | 17
pg/mL | -32 (28) | 66 (29) | 32 (26)

ADVERSE EVENTS:
Time Frame: throughout patient participation period of 8hr and up to 72 hrs follow-up after the dose administration
Description: No adverse events occurred during the study.
Arm/Group | Liraglutide 1.8 mg | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/17 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes